CLINICAL TRIAL: NCT05343481
Title: A Phase 2b, Open-label Study to Evaluate the Efficacy, Safety, Tolerability, Immunogenicity and Treatment Regimens of VTP-300 Combined With Low-dose Nivolumab in Chronic Hepatitis B Infection
Brief Title: Efficacy of VTP-300 in Chronic Hepatitis B Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBV-003
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B
Keywords: HBV, Chronic Hep B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Nivolumab; Solutions

STUDY DESIGN:
Intervention Model Description: Participants are randomised to the three treatment groups. Allocation to the groups is 1:1:1 allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Group 1 ChAdOx1-HBV, MVA-HBV and nivolumab (Experimental): Day 1: ChAdOx1-HBV 1 x 2.5 10^10 vp IM injection Day 29: MVA-HBV 1 x 10^8 pfu IM injection + nivolumab 0.3 mg/kg IV infusion
  Interventions: Biological: ChAdOx1-HBV; Biological: MVA-HBV; Biological: Nivolumab
- Experimental: Group 2 ChAdOx1-HBV, MVA-HBV and nivolumab, MVA-HBV and nivolumab (Experimental): Day 1: ChAdOx1-HBV 1 x 2.5 10^10 vp IM injection Day 29: MVA-HBV 1 x 10^8 pfu IM injection + nivolumab 0.3 mg/kg IV infusion Day 85: MVA-HBV 1 x 10^8 pfu IM injection + nivolumab 0.3 mg/kg IV infusion
  Interventions: Biological: ChAdOx1-HBV; Biological: MVA-HBV; Biological: Nivolumab
- Experimental: Group 3 ChAdOx1-HBV, MVA-HBV, nivolumab, MVA-HBV (Experimental): Day 1: ChAdOx1-HBV 1 x 2.5 10^10 vp IM injection Day 29: MVA-HBV 1 x 10^8 pfu IM injection Day 36: Nivolumab 0.3 mg/kg IV infusion Day 85: MVA-HBV 1 x 10^8 pfu IM injection
  Interventions: Biological: ChAdOx1-HBV; Biological: MVA-HBV; Biological: Nivolumab

INTERVENTIONS:
Biological: ChAdOx1-HBV — Chimpanzee Adenovirus Oxford 1-vectored Hepatitis B virus immunotherapeutic
Biological: MVA-HBV — Modified Vaccinia Ankara-vectored Hepatitis B virus immunotherapeutic
Biological: Nivolumab — Human immunoglobulin G4 monoclonal antibody
  Other Names: Opdivo 10mg/ml concentrate for solution for infusion

SUMMARY:
This is an open-label study to determine the efficacy, safety, tolerability and immunogenicity of ChAdOx1-HBV and MVA-HBV, together VTP-300, in combination with low-dose nivolumab, in patients with chronic HBV who are virally suppressed with oral anti-viral therapies.

DETAILED DESCRIPTION:
This is a multi-centre study conducted in 120 participants. All treatment groups will receive ChAdOx1-HBV on Day 1 and MVA-HBV on Day 29, and MVA boosts and nivolumab infusions as per treatment group as follows: Group 1: ChAdOx1-HBV, MVA-HBV and low dose nivolumab. Group 2: ChAdOx1-HBV, MVA HBV + low dose nivolumab, MVA HBV and low dose nivolumab. Group 3: ChAdOx1-HBV, MVA HBV, low dose nivolumab , MVA HBV. All participants return 7 days after each treatment (both immunotherapeutic and nivolumab infusion) visit to have chemistry and haematology safety laboratory studies obtained.

Participants are randomised to treatment in a 1:1:1 allocation. The primary objective of the study is to assess the efficacy of VTP-300 in combination with low-dose nivolumab in well-controlled CHB infection. The secondary objective of the study is to determine the safety and reactogenicity of the treatment regimens; this will be assessed by analysis of the incidence and severity of (serious) adverse events and any changes in laboratory values and vital signs. To assess the effect of VTP-300 in combination with low-dose nivolumab on the clearance of HBsAg and the impact of multiple booster doses of MVA-HBV and assess the appropriate timing of the use of low-dose nivolumab when used in combination with VTP-300.

Participants remain in the study for 12 months and attend clinic visits for treatment and assessments on Days 1, 8, 29, 36, 57, 85, 92, 113, 169, 252 and 336 (per Group allocation).

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged ≥18 to ≤65 years at screening (according to country/local regulations)
2. BMI ≤35 kg/m2
3. Able to provide informed consent indicating they understand the purpose of, and procedures required, for the study and are willing to participate
4. If female, willing not to become pregnant up to 8 weeks after the last dose of study vaccine and up to 5 months after the last dose of nivolumab
5. If female: Not pregnant or breast feeding and one of the following:

   * Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in ≥1 year and without an alternative medical cause)
   * Of childbearing potential but agrees to practice highly effective contraception for 4 weeks prior to study vaccine and 8 weeks after VTP-300 and 5 months after the last dose of nivolumab. Highly effective methods of contraception include one or more of the following:

     * Male partner who is sterile (medically effective vasectomy) prior to the female participant's entry into the study and is the sole sexual partner for the female participant
     * Combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal or transdermal
     * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable or implantable
     * An intrauterine device
     * Bilateral tubal occlusion
     * Abstinence from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent
6. Documented evidence of CHB infection (e.g., HBsAg positive ≥6 months with detectable HBsAg levels at screening; both HBeAg+ and HBeAg- allowed)
7. Receipt of only either entecavir, tenofovir (tenofovir alafenamide fumarate or tenofovir disoproxil fumarate) or besifovir for at least 6 months before screening
8. HBV-DNA viral load ≤ 1,000 IU/mL
9. HBsAg levels > 10 and ≤ 4,000 IU/mL

Exclusion Criteria:

1. Presence of any significant acute or chronic, uncontrolled medical or psychiatric illness in the opinion of the investigator would affect the safety of the participant or the evaluation of the data or interfere with adherence to the study requirements
2. Medical history that is thought to increase the participant's risk of reaction to a vaccine, including but not limited to capillary leak syndrome; transverse myelitis, Guillain Barré syndrome, thrombosis with thrombocytopenia syndrome (also termed vaccine-induced thrombotic thrombocytopenia); heparin-induced thrombocytopenia HCV RNA positive
3. HIV antibody positive and active hepatitis C (antibody positive and then DNA positive)
4. Co-infection with hepatitis D virus (HDV)
5. Documented cirrhosis or advanced fibrosis indicated by a liver biopsy within 6 months prior to Day 0 (Metavir activity grade A4 and stage F4; Ishak stages 5 - 6).
6. In the absence of a documented liver biopsy, either 1 of the following (not both):

   * Screening Fibroscan with a result >9 kilopascals (kPa) (or the equivalent) within ≤ 6 months of screening, OR
   * Both screening FibroTest >0.48 and aspartate aminotransferase (AST) to platelet ratio index (APRI) of >1.
7. ALT >3 x ULN, or INR >1.5 unless the participant was stable on an anticoagulant regimen affecting INR, albumin <3.2 g/dL, direct bilirubin >1.5 x ULN, platelet count <100,000/µL.
8. A history of liver decompensation (e.g., ascites, encephalopathy or variceal haemorrhage)
9. Prior hepatocellular carcinoma
10. Chronic liver disease of a non-HBV aetiology. (Note that Gilbert's syndrome, asymptomatic gallstones and non-alcoholic fatty liver not associated with steatohepatitis are not exclusions)
11. History or evidence of autoimmune disease or known immunodeficiency of any cause except history of autoimmune thyroiditis if the participant is stable on replacement therapy
12. Evidence of interstitial lung disease, active pneumonitis, myocarditis or a history of myocarditis
13. Prolonged therapy with immunomodulators (e.g., corticosteroids such as prednisone >10 mg/day) or biologics (e.g., monoclonal antibodies, IFN) within 3 months of Day 1. Inhaled, intra-articular, intra-bursal or topical corticosteroids are allowed. Physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed.
14. Receipt of immunoglobulin or other blood products within 3 months prior to Day 1
15. Receipt of any investigational drug or vaccine within 3 months prior to Day 1
16. Receipt of any non-oral adenoviral-based vaccine within 3 months prior to administration of ChAdOx1-HBV on Day 1
17. Severe reaction to any vaccine, requiring medical attention
18. Receipt of any live vaccines within 30 days prior to Day 1
19. Receipt of any inactivated non-live vaccines (e.g., mRNA, inactivated vaccines, toxoid vaccines) within 14 days prior to Day 1
20. History of severe hypersensitivity or anaphylactic reactions likely to be exacerbated by any component of VTP-300 or nivolumab, including severe allergy to egg
21. Malignancy within 5 years prior to screening with the exception of basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years. Participants under evaluation for possible malignancy are not eligible
22. Current alcohol or substance abuse judged by the investigator to potentially interfere with participant safety or compliance
23. Any laboratory test which is abnormal, and which is deemed by the investigator to be clinically significant
24. Any other finding that, in the opinion of the investigator, deems the participant unsuitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of participants with a greater than 1 log HBsAg | 6 months after the initiation of therapy
  Percentage of participants with a greater than 1 log HBsAg reduction at 6 months after initiation of therapy

SECONDARY OUTCOMES:
The incidence of participants with Treatment-Emergent Adverse Events (TEAEs) and ≥Grade 3 related adverse events following study treatment | From each study vaccination for the following 7 days
  The incidence of TEAEs and and ≥Grade 3 related adverse events will be based on the number and percentage of participants with events and number of events.
  TEAEs are defined as all adverse events occurring after study IMP administration; they will be further categorised by Seriousness, Severity (i.e. ≥ Grade 3) and Causality.
The incidence of participants with Treatment-Emergent Adverse Events (TEAEs) and ≥Grade 3 related adverse events following administration with nivolumab | From each study administration with nivolumab for the following 7days
  The incidence of TEAEs and ≥Grade 3 related adverse events will be based on the number and percentage of participants with events and number of events.
  TEAEs are defined as all adverse events occurring after study IMP administration with nivolumab; they are further categorised by Seriousness, Severity (i.e. ≥ Grade 3) according to FDA Guidance 70 FR 22664 and Causality.
The incidence of participants with Adverse Events of Special Interest (AESIs) | From study admission (the signature of informed consent) to the end of the study (Month 12)
  AESIs specific to this study include pneumonitis, grade 3 or 4 diarrhoea, diabetes, thyroid diseases, colitis, nephritis, immune-related endocrinopathies, myocarditis, immune-related skin conditions, or other unspecified immune-related adverse reactions
The incidence of participants with Treatment-Emergent Adverse Events (TEAEs) within each study group | From each study administration for the following 7 days
  The incidence of TEAEs will be based on the number and proportion of participants with events and number of events and will be calculated for each of the three study groups
Incidence of participants with potentially clinically significant laboratory signs within each treatment group as assessed by the Investigator | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  The incidence of participants will be based upon the number and proportion of patients in each treatment group with clinically significant laboratory signs (haematology and biochemistry, including liver function tests) as assessed by the investigator.
  All laboratory signs will be reported in SI units. If any laboratory sign is considered to be clinically significant i.e. outside laboratory normal reference range, the severity of this sign will be assessed according to the FDA Guidance for Industry 70 FR 22664. Absolute change, change from baseline and worst change for each participant will be calculated.
  The incidence of participants with treatment-emergent, clinically significant laboratory signs and laboratory signs of Grade 3-4 severity will be calculated for each treatment group at each time point
Incidence of participants with potentially clinically significant vital signs within each treatment group as assessed by the Investigator | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  The incidence of participants will be based upon the number and proportion of patients in each treatment group with clinically significant vital signs.
  Vital signs will be considered to be potentially clinically significant if they respectively fall below or above the relevant upper and lower limits.
  The incidence of participants with treatment-emergent, clinically significant vital signs will be calculated for each treatment group at each time point.
Number of participants with worst changes from baseline in laboratory hematology parameters | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  Hematology laboratory values will be evaluated according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA).
  For all hematology parameters, changes from baseline of at least two severity grades will be calculated for each timepoint at which the laboratory test is conducted throughout the study.
  The number of participants showing shifts of at least two severity grades (as worst change from baseline for each hematology parameter) will be presented within shift tables.
Number of participants with worst changes from baseline in laboratory biochemistry parameters | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  Biochemistry laboratory values will be evaluated according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA).
  For all biochemistry parameters, changes from baseline of at least two severity grades will be calculated for each timepoint at which the laboratory test is conducted throughout the study.
  The number of participants showing shifts of at least two severity grades (as worst change from baseline for each biochemistry parameter) will be presented within shift tables.
Number of participants with worst changes from baseline in laboratory urinalysis parameters | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  Urinalysis laboratory values will be evaluated according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA).
  For all urinalysis parameters, changes from baseline of at least two severity grades will be calculated for each timepoint at which the laboratory test is conducted throughout the study.
  The number of participants showing shifts of at least two severity grades (as worst change from baseline for each urinalysis parameter) will be presented within shift tables.
Number of participants with worst changes from baseline in vital signs parameters (heart rate, systolic blood pressure, diastolic blood pressure and temperature) | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  Worst change is defined as the lowest and highest post-baseline values for heart rate (bradycardia, tachycardia) and systolic blood pressure (hypotension, hypertension), and as the highest post-baseline values for diastolic blood pressure (hypertension) and temperature (fever).
  For all vital signs' measurements, changes from baseline will be calculated for each timepoint at which the vital sign measurement is conducted throughout the study. The number of participants showing worst change from baseline for the vital signs parameters overall will be presented within shift tables.
T cell response to the HBV antigen inserts of VTP-300 as measured by interferon (IFN)-γ enzyme-linked immunospot (ELISpot) | Baseline, Day 8, Day 29, Day 36, Day 57, Day 85, Day 92, Day 113, Day 169, Day 252 and Day 336
  This will be determined by using PMBCs in IFN-γ ELISpot assays to investigate the breadth of HBV specific T cell responses (defined by number of peptide pools or individual peptides recognised). These data may be used to build immunologic models of the immune system.

CONTACTS AND LOCATIONS:
Locations (18):
- Hong Kong (2):
  - Prince Of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Taiwan (8):
  - Chia-Yi Christian Hospital, Chiayi City
  - Dalin Tzu Chi Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (8):
  - Chulabhorn Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - HIV Netherlands-Australia-Thailand Research Collaboration, Bangkok
  - Hospital For Tropical Diseases, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Research Institute For Health Sciences, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi

IPD SHARING:
Plan to Share IPD: No